CLINICAL TRIAL: NCT07376083
Title: Comparison of the Diagnostic Accuracy of Bedside Gastric Ultrasonography and Chest Radiography for Verification of Nasogastric Feeding Tube Placement in Intensive Care Unit Patients: A Prospective Observational Study
Brief Title: Ultrasound vs Chest X-ray for NG Tube Placement in ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Guldem Turan, Prof., Tepecik Training and Research Hospital
Other Study IDs: 2025/11-04
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Intensive Care (ICU)
Keywords: Nasogastric Tube Placement, Point-of-Care Ultrasonography, Diagnostic Accuracy Chest X-ray , Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
his study evaluates the diagnostic accuracy of bedside gastric ultrasonography for confirmation of nasogastric tube placement in intensive care unit patients, using chest radiography as the reference standard. Sensitivity and specificity of bedside ultrasonography will be calculated to assess its performance in this clinical setting.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Clinical indication for nasogastric tube placement

Written informed consent obtained from the patient or a legally authorized representative

Exclusion Criteria:

* Refusal to participate in the study

Age < 18 years

Pregnancy

Contraindications to nasogastric tube placement, including:

Facial trauma

Basilar skull fracture

Esophageal obstruction

Recent upper gastrointestinal surgery

Presence of wounds, burns, or surgical dressings in the epigastric region that preclude adequate ultrasonographic evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 years and older) admitted to the intensive care unit who have a clinical indication for nasogastric tube placement. Eligible patients are enrolled prospectively following written informed consent obtained from the patient or a legally authorized representative.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of bedside gastric ultrasonography for confirmation of nasogastric tube placement | Immediately after nasogastric tube placement
  Diagnostic accuracy of bedside gastric ultrasonography will be assessed by calculating sensitivity and specificity using chest radiography as the reference standard.

SECONDARY OUTCOMES:
Agreement between bedside gastric ultrasonography and chest radiography | Immediately after nasogastric tube placement
  The level of agreement between bedside gastric ultrasonography and chest radiography findings will be evaluated.
Time to confirmation of nasogastric tube placement | From tube insertion to confirmation
  Time required to confirm correct nasogastric tube placement using bedside gastric ultrasonography and chest radiography.

IPD SHARING:
Plan to Share IPD: No